CLINICAL TRIAL: NCT05265494
Title: Let´s Talk About Sleep in College Student: an Innovative Treatment Based on Non-invasive Neuromodulation to Enhance the Sleep Quality and Academic Efficiency: Randomised Controlled Trial" (USLEEP)
Brief Title: Let´s Talk About Sleep in College Student
Acronym: USLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Collaborators: Alfonso X El Sabio University (Other); University of Alcala (Other); University Pontifical of Salamanca (Unknown)
Responsible Party: Principal Investigator, Daniel David Álamo Arce, Principal Investigator, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USLEEP; 001 (Other: ULPGC)
Record Dates: First submitted 2021-11-05; First posted 2022-03-03 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Stress; Sleep Disturbance
Keywords: sleep; neuromodulation; academic performance; students
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with passive control, triple blind (for the patient, the physiotherapist applying the technique and evaluator), with a parallel and multicenter design. The study will have two arms or groups; the intervention group (G1) will undergo neuromodulation treatment with the NESA XSIGNAL® device and the control group (G2) will not carry out any intervention, but both will be evaluated for the same variables at the same times.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The intervention to which the subjects have been assigned, the specialist and the researcher who collects the information and carries out the follow-ups will be blinded. Data analysis will also be performed in a blinded way.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NESA INTERVENTION (Experimental): Group 1: Application of Nesa microcurrents through the NXSIGNAL® generator twice a week.
  The study volunteers are treated with the NXSIGNAL® device in sessions of 60 minutes, twice a week and for 5 weeks (10 sessions).
  Interventions: Device: Non invasive neuromodulation NESA (XSIGNAL device)
- CONTROL-NO INTERVENTION (No Intervention): Group 2: Control group without NESA XSIGNAL® application The same protocol for the analysis of variables is followed, but without performing any type of treatment with the NESA XSIGNAL device.

INTERVENTIONS:
Device: Non invasive neuromodulation NESA (XSIGNAL device) — The study volunteers are treated with the NXSIGNAL® device in sessions of 60 minutes, twice a week and for 5 weeks (10 sessions).
  • The skin must be clean, free of creams and grease, lectrodes are connected to the control console and the targeting electrode located in over the intervertebral area between C7 and T1 (cervical area) and will follow the central treatment pattern with the following combination:
  * 2 sessions: Program 1 (30 min), Program 7 (15min) and Program 8 (15min).
  * 4 sessions: Program 2 (15min), Program 7 (30 min) and Program 8 (15min)
  * 4 sessions: Program 7 (60min)
  Arms: NESA INTERVENTION

SUMMARY:
The concern about the quality of sleep of university students, future professionals of the world, must be crucial for the scientific community, as well as for university professors and professors. Innovative electrotherapy technologies such as non-invasive neuromodulation NESA are demonstrating effects on improving sleep quality, concentration and stress, so the objective of this project is to carry out a triple-blind randomized clinical trial with first-year science science students. health from three universities. The design is made up of an intervention group with NESA technology and another control group in each of the centers. Where the quality of sleep, perception of stress, cortisol levels in saliva and academic performance will be analyzed.

This multicenter project hopes to demonstrate that non-invasive NESA neuromodulation can be a preventive treatment for the maintenance of sleep quality during stressful periods such as university exams, as well as being able to modulate perceived stress and translate into an improvement in student performance.

DETAILED DESCRIPTION:
Randomized clinical trial with passive control, triple-blind, with a parallel and multicenter design. The study will have two arms; the intervention group will have neuromodulation treatment with the NESA XSIGNAL® device and the control group will not carry out any intervention, but both will be evaluated for the same variables at the same times.

Multicenter study whose collaborating entities correspond to the University of Las Palmas de Gran Canaria, Alfonso X el Sabio University, the Pontifical University of Salamanca and the University of Alcalá de Henares. The study population will be students from the collaborating universities, corresponding to first-year health sciences degrees. For the selection of the sample, a non-probabilistic convenience sampling will be carried out, which allows selecting those accessible cases that agree to be included.

Patients who agree to participate will be randomly assigned to one of the 2 arms of the study (real device or control), using a fixed-size block design generated by the data manager to guarantee balanced randomization for each of the arms and in each of the participating universities. The assignment process will be carried out hidden and will be carried out by the support researcher in the Unit indicated for this study. Each research subject will be assigned an identification code corresponding to correlative numbers from 1 to 80, being from 1-20 subjects of the UPSA, from 21-40 students of the Alfonso X el Sabio University, from 41 to 60 students from the University of Las Palmas and from 61 to 80 from the University of Alcalá.

The intervention to which the subjects have been assigned, the specialist and the researcher who collects the information and carries out the follow-ups will be blinded. Data analysis will also be performed in a blinded fashion.

The default schedule is based on the goals set in this study. The main goal is to improve the quality of sleep. The secondary objectives are to correlate with improving the perception of stress and academic performance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people
* Be enrolled in a degree in health sciences at the partner universities in the study in the first year.
* Optimal cognitive abilities and mentally competent to participate in the study.
* In cognitive conditions to complete the study questionnaires
* Have an optimal command of the Spanish language to complete the questionnaires.
* Signing of the informed consent for participation

Exclusion Criteria:

* Present some of the contraindications for a treatment with NESA XSIGNAL®: Pacemaker or other electrical surgical device, internal bleeding, do not apply electrodes on skin in poor condition, with ulcerations or wounds, acute febrile processes, pregnancy, acute thrombophlebitis and / or phobia to electricity, and pregnant.
* Combine another pharmacological treatment that influences the variables to be evaluated during the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Sleep quality | At the first consultation and through study completion, 5 weeks
  Through a validated sleep quality perception questionnaire, Pittsburgh questionnaire. the Pittsburgh index scored by the higher the total score, the worse the quality of sleep. In this way, a total score less than or equal to five indicates that, in general, your quality of sleep is optimal, while a total score greater than five suggests that you have more or less serious sleep problems.
Salival Cortisol | At the first consultation and through study completion, 5 weeks
  Through the Soma OFC II cube. The analysis will be performed in real time through the collection of saliva, it is not affected by recent food and drink; Once the swab is in the buffer, your sample is stable for months. It is a validated instrument

SECONDARY OUTCOMES:
Academic Stress | At the first consultation and through study completion, 5 weeks
  The questionnaire Academic Stress Questionnaire at University (Time Management Behavior Questionnaire for University Students, in english). It assesses possible stressful situations in the university environment and consists of a total of 21 items. The participants' responses indicate the level of perceived stress in each situation using a Likert-type response scale with 5 options ranging from "no stress" (1) to "a lot of stress" (5). .
  The scale evaluates four complementary dimensions:
  * Establishing objectives and priorities. Its response range lies between 10-50, and its internal consistency is .90.
  * Time management tools. A response range between 11-55 and an internal consistency of .88.
  * Preferences for disorganization. A response range between 8-40 and an internal consistency of .70.
  * Perception of control over time. A response range between 5-25 and an internal consistency of .68
Coping with academic stress | At the first consultation and through study completion, 5 weeks
  The Academic stress coping scale, known as A-CEA (Escala de afrontamiento del estrés académico, in spanish) (González Cabanach et al., 2010), is a subscale of the CEAU questionnaire. It evaluates the establishment of adequate time periods for studying (daily, weekly, monthly), the effective use of time, setting realistic objectives, and the characteristics of the setting in which the subject usually studies and does his or her academic activities. It consists of 8 items (e.g., "I make sure I am caught up on the material and projects"), with a response range between 8-56 and an internal consistency of .79.
Questionnaire of sociodemographic variables | At the first consultation and through study completion, 5 weeks
  A third questionnaire to collect necessary information on sociodemographic variables such as age, gender, place of residence and type of home. This questionnaire also aims to collect some data regarding their academic life, such as the average grade for access to university and the degree completed. The ad-hoc questionnaire consists of a total of 11 items and all questions are made in a clear and concise manner so that the answer is free from ambiguity.
ACADEMIC PERFORMANCE | Through study completion, 5 weeks
  The final average grade of the first academic semester will be analyzed comparing by groups.

CONTACTS AND LOCATIONS:
Overall Officials: Raque l I Medina Ramírez, PhD, Study Director — University of Las Palmas de Gran Canaria
Locations (2):
- Spain (2):
  - Raquel Irina Medina Ramirez, Las Palmas de Gran Canaria, Las Palmas
  - María Miana, Madrid

IPD SHARING:
Plan to Share IPD: No
All data will be collected by computer in an encrypted Excel document (Microsoft Office Excel 2019 MSO 64-bit program).
  Everything is collected in accordance with the provisions of Organic Law 3/2018, of December 5, on the Protection of Personal Data and guarantee of digital rights and by virtue of the provisions of Regulation (EU) 2016/679 of the European Parliament and of the Council, of April 27, 2016, regarding the protection of natural persons with regard to the processing of personal data and the free circulation of these data.

REFERENCES:
- [Background] Gaultney JF. The prevalence of sleep disorders in college students: impact on academic performance. J Am Coll Health. 2010;59(2):91-7. doi: 10.1080/07448481.2010.483708. PMID 20864434
- [Background] Escobar-Cordoba F, Eslava-Schmalbach J. [Colombian validation of the Pittsburgh Sleep Quality Index]. Rev Neurol. 2005 Feb 1-15;40(3):150-5. Spanish. PMID 15750899

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT05265494/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT05265494/ICF_001.pdf